CLINICAL TRIAL: NCT04684602
Title: Evaluation of the Safety, Tolerability and Efficacy of Regenerative Therapy for the Treatment of Various Chronic and Acute Conditions
Brief Title: Mesenchymal Stem Cells for the Treatment of Various Chronic and Acute Conditions
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Advanced Medical LLC (Industry)
Collaborators: HeartStem Institute (Unknown); NuStem (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICSS-2020-032
Record Dates: First submitted 2020-12-02; First posted 2020-12-24 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Autoimmune Diseases; Cardiovascular Disorders; Diabetes Complications; Integumentary Disease; Musculoskeletal Disorders; Neurodegenerative Disorders; Neurologic Disorders; Pulmonary Disorders; Sexual Dysfunction; Urologic Disorders; Viral Illness
Keywords: stem cell therapy; umbilical cord stem cells; amniotic stem cells; stem cells; MSC; Mesenchymal Stem Cell; Medicinal Signaling Cell; Erectile Dysfunction; Heart Diseases; Mental Disorders; Neurocognitive Disorders; Neurodegenerative Diseases; Central Nervous System Diseases; Tauopathies; Brain Diseases; Dementia; Disease; Cardiomyopathies; Urologic Diseases; Peripheral Nervous System Diseases; Nervous System Diseases; Alzheimer Disease; Musculoskeletal Diseases; Cardiovascular Diseases; Immune System Diseases; Neuromuscular Diseases; Covid-19
MeSH Terms: conditions — Autoimmune Diseases; Cardiovascular Diseases; Diabetes Complications; Skin Diseases; Musculoskeletal Diseases; Neurodegenerative Diseases; Nervous System Diseases; Lung Diseases; Sexual Dysfunction, Physiological; Urologic Diseases; Virus Diseases; Erectile Dysfunction; Heart Diseases; Mental Disorders; Neurocognitive Disorders; Central Nervous System Diseases; Tauopathies; Brain Diseases; Dementia; Disease; Cardiomyopathies; Peripheral Nervous System Diseases; Alzheimer Disease; Immune System Diseases; Neuromuscular Diseases; COVID-19

STUDY DESIGN:
Intervention Model Description: This is a multi-center, prospective, open label clinical trial. It will include 5000 patients suffering acute and chronic conditions under 10 different categories. Patients will undergo a single treatment with a biological tissue allograft and will be followed for 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (10):
- Arm 1: Autoimmune Diseases (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for autoimmune conditions. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 2: Cardiovascular Disorders (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for cardiovascular disorders and conditions. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 3: Diabetes Complications (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for diabetes complications. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 4: Integumentary Disease (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for integumentary diseases and conditions. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 5: Musculoskeletal Disorders (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for orthopedic and musculoskeletal conditions. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 6: Neurodegenerative Disorders (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for neurologic and neurodegenerative disorders. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 7: Pulmonary Disorders (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for pulmonary disorders. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 8: Sexual Dysfunction (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for sexual dysfunction conditions. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 9: Urologic Disorders (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for urologic conditions. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™
- Arm 10: Viral Illnesses (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for viral illnesses. Outcomes will be compared to results in peer-reviewed literature for several conditions.
  Interventions: Biological: PrimePro™/ PrimeMSK™

INTERVENTIONS:
Biological: PrimePro™/ PrimeMSK™ — Injection via condition specific route of administration.

SUMMARY:
This multi-arm, multi-site study investigates the safety, tolerability, and efficacy of stem cell therapy for the treatment of various acute and chronic conditions. Clinically observed initial findings and an extensive body of research indicate regenerative treatments are both safe and effective for the treatment of multiple conditions.

DETAILED DESCRIPTION:
This multi-arm, multi-site study investigates the safety, tolerability, and efficacy of stem cell therapy for the treatment of various acute and chronic conditions. Clinically observed initial findings and an extensive body of research indicate regenerative treatments are both safe and effective for the treatment of multiple conditions.

This study investigates clinical outcomes of treatments for numerous indications including: Autoimmune, Cardiovascular, Diabetes, Integumentary, Neurologic / Neurodegenerative, Pulmonary, Orthopedic Diseases, Sexual Dysfunction, Urologic Disorders and Viral Illnesses.

Our hypotheses posit that regenerative treatments are both safe and statistically beneficial for a range of conditions. Outcomes will be determined by multiple valid outcome instruments that measure general quality of life information along with condition-specific information.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Ability to provide informed consent
* Availability for follow up visits

Exclusion Criteria:

* Active or recent malignancy (within last 2 years)
* Pregnancy or breast-feeding
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2030-07-09 (Estimated); Study Completion 2030-12-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of quality of life (QOL) via 36-Item Short Form Survey (SF-36) change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  General Health Outcome Instrument used to derive a simple psychometric score for health related quality of life which provides scores on various dimensions or items describing the systems. The score is derived by adding the unweighted response order of each question, with a lower score denoting a better quality of life.
Assessment of disabilities of arm, shoulder, hand via DASH Questionnaire change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  Upper Extremity Outcome Instrument
Assessment of erectile function via International Index of Erectile Function (IIEF-5) change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  Erectile Function Questionnaire. Scoring exists from 0 to 25. The lower the score, the more severe the Erectile Dysfunction.
Assessment of COPD via Clinical Chronic Obstructive Pulmonary Disease Questionnaire change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  COPD Outcome Instrument. Items are scored on a Likert scale (range 0-60). Higher scores indicate a worse health status.
Assessment of mental state via Mini Mental State Examination (MMSE) change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  Memory Outcome Instrument. The maximum MMSE score is 30 points. The lower the score, the more severe the dementia.
Assessment of interstitial cystitis via O'Leary/Sant Questionnaire change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  Voiding and Pain Indices. Possible score of 0-20 with higher scores denoting better function.
Assessment of back pain via Oswestry Low Back Pain Disability Questionnaire change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  Low Back Pain Outcome Instrument. Possible score of 0-100 with lower scores denoting better function.
Assessment of osteoarthritis via Western Ontario and McMaster Osteoarthritis Index (WOMAC) change from baseline at 6 and 12 months. | Follow up time-frames will measure changes occurring from baseline post procedure at 6 months and 12 months.
  Arthritis Outcome Instrument. Individual question scores are then summed to form a raw score ranging from 0 (worst) to 96 (best)

CONTACTS AND LOCATIONS:
Overall Officials: Ernst R Von Schwarz, MD, PhD, Principal Investigator — HeartStem Institute, Southern California Hospital at Culver City
Locations (1):
- Southern California Hospital at Culver City / Southern California Hospital at Hollywood / Multiple US-based Sub-Investigator Sites, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will be blinded and password protected. Research publications will be produced for medical journals. Participating Investigators will have password protected access only.